CLINICAL TRIAL: NCT03763526
Title: Association Between Perioperative Nutritional Status and Surgical Outcome in Digestive System Cancer Patients
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/526
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Digestive System Cancer
Keywords: Perioperative Nutritional Status; Surgical Outcome in Digestive System Cancer
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Malnutrition is a common problem in cancer patients. It negatively inﬂuences patients' prognosis and quality of life. In gastrointestinal patients, it is also caused by insufﬁcient food intake due to dysphagia, lack of appetite, nausea, vomiting, impaired digestion and absorption.

Furthermore, influence of prior oncologic treatment (surgery, chemotherapy, and radiotherapy), have been associated with prolonged hospital stay, more postoperative complications and low survival outcome1-4. So, the proper assessment of nutrition status to detect perioperative malnutrition may allow appropriate nutritional therapy and improve survival5.

However, the important factor which prolongs survival rate is good preoperative nutrition status because it effects the postoperative nutrition outcome. The objective of this study is to correlate the association between pre- and postoperative nutrition status and surgical outcomes.

The Nutrition Alert Form (NAF) is a clinical tool for determining nutritional status. The NAF was modified from Subjective Global Assessment (SGA)6, and it is easy to use and does not require nutritional expertise based on laboratory and physical examination. Therefore, the NAF has been used extensively for screening of malnutrition in hospitalized Thai patients and it can classify the nutritional status into three groups : NAF-A (Normal-Mild malnutrition), NAF-B (Moderate malnutrition), NAF-C (Severe malnutrition)

DETAILED DESCRIPTION:
Primary Questions

- What is the relationship between the preoperative nutrition status and the postoperative nutrition status in gastrointestinal cancer patients ?

Secondary Questions

- What is the relationship between malnutrition during preoperative and postoperative stages, compared with postoperative complications?

OBJECTIVE :

The objective of this study is to study the association between pre- and postoperative nutrition status compared with postoperative complications and surgical outcome. The results of this study may affect future nutrition practices and encourage different behaviors in gastrointestinal cancer patients who prepare to undergo surgery.

Sample size is calculated by n=(z_(1-α/2)^2 p(1-p))/d^2

Proportion (p) = 0.80, Error (d) = 0.064 Alpha (α) = 0.05, Z(0.975) = 1.959964 Power = 0.80 Sample size (n) = 178 Include drop out 10 % = 196 patients

Patients:

For 196 gastrointestinal cancer patients (esophageal, gastric, colon and rectum cancer), who underwent scheduled surgery. Every patient underwent nutritional assessment by NAF before surgery and (1 & 3 months) after surgery at in the Department of Surgery, Ramathibodi Hospital and Buriram Hospital from 20 November 2018. Patients with incomplete documents were excluded from this study.

DATA COLLECTION AND DATA ANALYSIS:

* Pre-operative nutrition status assess by NAF
* Post-operative nutrition status at 1 month and 3 months assess by NAF
* All postoperative complications were collected according to Clavin-Dindo Classification8
* All case were included in this study, following TNM staging and others pathologic parameters :
* Cancer type - Tumor grading
* Lymph node metastasis - Tumor depth

ELIGIBILITY:
Inclusion Criteria:

* All patients GI cancer
* Elective surgery

Exclusion Criteria:

* Lack of oncologic treatment information before surgery
* No history of recurrent cancer or more than one cancer disease
* Patients who have been diagnosed with Carcinomatosis peritonei during the operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: gastrointestinal cancer patients (esophageal, gastric, colon and rectum cancer), who underwent scheduled surgery.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 1 month
  The complication were collected according to Clavin-Dindo Classification
postoperative complications | 3 month
  The complication were collected according to Clavin-Dindo Classification

SECONDARY OUTCOMES:
operative nutrition status | 1 month
  operative nutrition status assess by Nutrition Alert Form (NAF)
operative nutrition status | 3 month
  operative nutrition assess by Nutrition Alert Form (NAF)

OTHER OUTCOMES:
Length of hospital stay | 1 month
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Supsamutchai, MD, Study Chair — Ramathibodi Hospital
Locations (1):
- Chairat Supsamutchai, Bangkok, Bankok, Thailand